CLINICAL TRIAL: NCT07323888
Title: Comparison of Traditional Radiofrequency Ablation of Inferior Turbinates With or Without Posterior Nasal Radiofrequency Ablation: A Randomized Controlled Trial
Brief Title: Traditional vs. Posterior Nasal Radiofrequency Ablation for Chronic Rhinitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chien Yu Huang (Other)
Responsible Party: Sponsor-Investigator, Chien Yu Huang, Attending Physician, Department of Otolaryngology, Chia-Yi Hospital, Ministry of Health and Welfare
Organization: Chia-Yi Hospital, Ministry of Health and Welfare (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 25-013; 25-013 (Other: Institutional Review Board, Jianan Psychiatric Center, MOHW)
Record Dates: First submitted 2025-12-12; First posted 2026-01-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Nasal Obstruction; Chronic Rhinitis; Nonallergic Rhinitis; Rhinorrhea; Inferior Turbinate Hypertrophy
Keywords: Radiofrequency Ablation; Inferior Turbinate Hypertrophy; Chronic Rhinitis; Nasal Obstruction; Rhinorrhea; Posterior Nasal Nerve; Randomized Controlled Trial; Single-Center Study
MeSH Terms: conditions — Nasal Obstruction; Rhinorrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferior Turbinate RF with Posterior Nasal RF Ablation (Experimental): Traditional Radiofrequency Ablation of Inferior Turbinates With Posterior Nasal Radiofrequency Ablation
  Interventions: Procedure: Traditional Radiofrequency Ablation of Inferior Turbinates With Posterior Nasal Radiofrequency Ablation
- Inferior Turbinate RF Ablation (Active Comparator): Traditional Radiofrequency Ablation of Inferior Turbinates
  Interventions: Procedure: Traditional Radiofrequency Ablation of Inferior Turbinates

INTERVENTIONS:
Procedure: Traditional Radiofrequency Ablation of Inferior Turbinates With Posterior Nasal Radiofrequency Ablation — Intervention:
  Radiofrequency Ablation (Olympus Celon Elite ESG-400)
  * Local anesthesia with 2% lidocaine
  * RF ablation at 15W
  * Multiple punctures along anterior, middle, and posterior inferior turbinate (15-20 per side)
  * Includes posterior nasal region (superior, medial, inferior aspects)
  * No nasal packing required
  Post-operative care (3 days):
  1. Tranexamic acid 250mg 1cap BID x3 days
  2. Amoxicillin 500mg 1 cap BID x3 days
  3. Acetaminophen 500mg 1tab BID x3 days
  4. Levocetirizine 5mg 1tab QD x3 days + PRN x4 days
  Arms: Inferior Turbinate RF with Posterior Nasal RF Ablation
Procedure: Traditional Radiofrequency Ablation of Inferior Turbinates — Intervention:
  Radiofrequency Ablation (anterior inferior turbinate only)
  * Same anesthesia and device
  * RF applied only to anterior inferior turbinate (≈2 punctures per side)
  * No treatment to middle/posterior inferior turbinate Post-operative care: Same as experimental arm
  Arms: Inferior Turbinate RF Ablation

SUMMARY:
This study is a prospective, single-center, single-blinded randomized controlled trial designed to compare the clinical effectiveness of traditional radiofrequency ablation of the anterior inferior turbinate alone versus expanded radiofrequency ablation including the middle and posterior portions of the inferior turbinate (posterior nasal region). Patients with chronic rhinitis who remain symptomatic despite at least six months of medical therapy will be randomized in a 2:1 ratio to undergo extended posterior nasal ablation versus traditional anterior treatment. Symptom improvement will be evaluated using rTNSS and other validated questionnaires.

DETAILED DESCRIPTION:
Chronic rhinitis is a common condition characterized by persistent nasal obstruction and rhinorrhea, leading to significant impairment in quality of life. Radiofrequency ablation of the inferior turbinate is an established minimally invasive treatment for patients with symptoms refractory to medical therapy. However, symptom control may be suboptimal in some patients, particularly when posterior nasal neural components contribute to disease persistence.

Posterior nasal radiofrequency ablation, which extends treatment to the middle and posterior portions of the inferior turbinate, has been proposed as an adjunctive technique to enhance symptom relief by targeting posterior nasal regions. Evidence comparing traditional anterior inferior turbinate radiofrequency ablation with expanded posterior nasal radiofrequency ablation remains limited.

In this prospective, single-center, randomized controlled trial, eligible patients with chronic rhinitis refractory to at least six months of medical therapy will be randomized in a 2:1 ratio to receive either expanded radiofrequency ablation including the middle and posterior portions of the inferior turbinate or traditional anterior inferior turbinate radiofrequency ablation alone. The primary outcome is the response rate based on improvement in reflective Total Nasal Symptom Score (rTNSS), defined as a ≥30% reduction from baseline at 3 months after the procedure. Secondary outcomes include changes in validated symptom and quality-of-life questionnaires and the incidence of procedure-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Chronic rhinitis symptoms for at least 6 months that have not responded effectively to medication (should include at least Intranasal corticosteroid (ICS) combined with intermittent use of oral antihistamine and, as needed, combination nasal spray) or where medication has not provided sustained improvement
* Total rTNSS ≥ 4 with Moderate to severe rhinorrhea symptoms (24-hour reflective Total Nasal Symptom Score [rTNSS] rhinorrhea score of 1-3) and mild to severe nasal congestion symptoms (rTNSS nasal congestion score of 1-3)
* All enrolled patients routinely undergo endonasal endoscopic examination, or have had a sinus CT within the past month confirming no significant rhinosinusitis."

Exclusion Criteria:

* Obstructive anatomical abnormalities limiting access to posterior nasal passages
* Nasal anatomical changes due to previous sinus or nasal surgery or injury
* Ongoing nasal or sinus infection
* History of severe dry eye, chronic epistaxis, rhinitis medicamentosa, or head and neck radiotherapy
* Self-reported history of bleeding tendency
* Current use of anticoagulants with inability to discontinue
* Previous chronic rhinitis surgery
* History of poor wound healing after head, neck, or throat surgery
* Pregnancy/lactation
* Neuromuscular disease preventing supine positioning

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Response rate based on improvement in reflective Total Nasal Symptom Score (rTNSS) | 3 months after the procedure
  Response is defined as a ≥30% reduction from baseline in the reflective Total Nasal Symptom Score (rTNSS; range 0-12, higher scores indicate worse symptoms).

SECONDARY OUTCOMES:
Change in reflective Total Nasal Symptom Score (rTNSS) | Baseline, 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months after the procedure
  Change in reflective Total Nasal Symptom Score (rTNSS; range 0-12, higher scores indicate worse symptoms) from baseline.
Change in Nasal Obstruction Symptom Evaluation (NOSE) score | Baseline, 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months after the procedure
  Change in Nasal Obstruction Symptom Evaluation (NOSE; range 0-20, higher scores indicate worse symptoms) from baseline.
Change in Mini Rhinoconjunctivitis Quality of Life Questionnaire (Mini-RQLQ) score | Baseline and 3 months after the procedure
  Change in Mini Rhinoconjunctivitis Quality of Life Questionnaire (Mini-RQLQ; range 0-6, higher scores indicate worse quality of life) from baseline.
Incidence of intervention-related complications | From the date of the procedure through 12 months after the procedure
  All self-reported and clinically observed complications related to the intervention.
Change in Eustachian Tube Dysfunction Questionnaire-7 (ETDQ-7) score | Baseline and 3 months after the procedure
  Change in Eustachian Tube Dysfunction Questionnaire-7 (ETDQ-7; range 7-49, higher scores indicate worse symptoms) from baseline.
Change in Patulous Eustachian tube handicap inventory-10 (PHI-10) score | Baseline and 3 months after the procedure
  Change in Patulous Eustachian tube handicap inventory-10 (PHI-10; range 0-40, higher scores indicate worse symptoms) from baseline.
Change in Pittsburgh Sleep Quality Index (PSQI) score | Baseline and 3 months after the procedure
  Change in Pittsburgh Sleep Quality Index (PSQI; range 0-21, higher scores indicate worse sleep quality) from baseline.
Change in Epworth Sleepiness Scale (ESS) score | Baseline and 3 months after the procedure
  Change in Epworth Sleepiness Scale (ESS; range 0-24, higher scores indicate greater daytime sleepiness) from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Chiayi Hospital, Ministry of Health and Welfare (MOHW), Chiayi City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient privacy considerations and institutional data protection policies. Only aggregated results will be presented in publications and reports.

REFERENCES:
- [Background] Stolovitzky JP, Ow RA, Silvers SL, Bikhazi NB, Johnson CD, Takashima M. Effect of Radiofrequency Neurolysis on the Symptoms of Chronic Rhinitis: A Randomized Controlled Trial. OTO Open. 2021 Sep 10;5(3):2473974X211041124. doi: 10.1177/2473974X211041124. eCollection 2021 Jul-Sep. PMID 34527852
- [Background] Ehmer D, McDuffie CM, Scurry WC Jr, McIntyre JB, Mehendale NH, Willis JH, Shealy RB, Watkins JP, Kakarlapudi VV. Temperature-Controlled Radiofrequency Neurolysis for the Treatment of Rhinitis. Am J Rhinol Allergy. 2022 Jan;36(1):149-156. doi: 10.1177/19458924211033400. Epub 2021 Aug 12. PMID 34382444
- [Background] Lee JT, Abbas GM, Charous DD, Cuevas PDMM, Goktas PDMO, Loftus PA, Nachlas NE, Toskala EM, Watkins JP, Brehmer PDMD. Clinical and Quality of Life Outcomes Following Temperature-Controlled Radiofrequency Neurolysis of the Posterior Nasal Nerve (RhinAer) for Treatment of Chronic Rhinitis. Am J Rhinol Allergy. 2022 Nov;36(6):747-754. doi: 10.1177/19458924221109987. Epub 2022 Jul 11. PMID 35818709
- [Background] Takashima M, Stolovitzky JP, Ow RA, Silvers SL, Bikhazi NB, Johnson CD. Temperature-controlled radiofrequency neurolysis for treatment of chronic rhinitis: 12-month outcomes after treatment in a randomized controlled trial. Int Forum Allergy Rhinol. 2023 Feb;13(2):107-115. doi: 10.1002/alr.23047. Epub 2022 Jul 5. PMID 35714267
- See also: Position Statement: PNN Ablation for the Treatment of Chronic Rhinitis — https://www.entnet.org/resource/position-statement-posterior-nasal-nerve/